CLINICAL TRIAL: NCT05731791
Title: A Prospective Randomized Trial to Compare MRI-guided Precision Prone Irradiation (PPI) Versus CT-guided Breast Irradiation
Brief Title: Trial to Compare MRI-guided Precision Prone Irradiation (PPI) Versus CT-guided Breast Irradiation
Acronym: PPI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-01024342
Record Dates: First submitted 2023-02-07; First posted 2023-02-16 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Phase 3 two-armed randomized clinical trial for localized favorable breast cancer patients, randomizing to CT-based radiation treatment vs. MRI-based radiation treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- ARM 1 - CT-based breast radiation treatment (Active Comparator): Patients randomized to ARM 1 will receive 3000 cGy in 5 fractions partial breast radiotherapy with CT-based breast radiation treatment.
  Interventions: Radiation: Radiation Therapy to partial breast
- ARM 2 - MRI-based breast radiation treatment (Active Comparator): Patients randomized to ARM 2 will receive 3000 cGy in 5 fractions partial breast radiotherapy with MRI-based breast radiation treatment.
  Interventions: Radiation: Radiation Therapy to partial breast

INTERVENTIONS:
Radiation: Radiation Therapy to partial breast — Patients randomized to ARM 1 will receive 3000 cGy in 5 fractions partial breast radiotherapy with CT-based breast radiation treatment (Arm 1) and patients randomized to ARM 2 will receive 3000 cGy in 5 fractions partial breast radiotherapy with MRI-based breast radiation treatment (Arm 2).

SUMMARY:
The Investigators are investigating the potential role of MRI-guided Radiation Therapy for patients receiving breast radiotherapy in the prone position with a MRI-Linac radiotherapy system, the Precision Prone Irradiation (PPI) technique.

Hypothesis: The investigators would like to hypothesize that breast radiation therapy using MRI-guided system including the MRI-Linac (Arm 2) is comparable to the current standard of treatment using conventional CT-based system (Arm 1), in terms of local control of the disease at 2 year time point.

DETAILED DESCRIPTION:
Breast conserving surgery and adjuvant whole breast radiotherapy is a standard treatment option for most patients with early-stage invasive breast cancer. Recent technological advances in radiotherapy have enabled shorter treatment courses, smaller radiation fields, prone positioning, and fewer side effects associated with breast cancer treatment. To further improve target accuracy in breast radiation delivery, an emerging radiotherapy technology takes advantage of on-table MRI imaging and daily adaptive planning during the radiation delivery process.

The objectives of the study are to compare side effects in patients treated under either of these treatment settings and to compare recurrence (if the cancer comes back) rates at a 2-year time point. Patients will have annual follow ups up to 10 years and recurrence rates will be measured at 5-year and at 10-year time points.

ELIGIBILITY:
Patients ≥ 50 yrs with histologically confirmed unilateral DCIS or Stage I invasive breast cancer; received breast conserving surgery (pN0 or pNx) with tumor pathology ≤ 2 cm and excision margin ≥ 1 mm

Inclusion Criteria:

* Women status post segmental mastectomy
* If unilateral, pT1 breast cancer excised with negative margins AND/OR pTis excised with negative margins.
* If bilateral, pT1 breast cancer excised with negative margins AND/OR pTis excised with negative margins.
* Clinically N0 or pN0 or sentinel node negative
* Ductal carcinoma in situ DCIS with negative margins (no DCIS on inked margins).

Exclusion Criteria:

* Previous radiation therapy to the ipsilateral breast.
* > 90 days from last surgery, unless s/p adjuvant chemotherapy
* > 60 days from last chemotherapy
* Patients unable to tolerate MRI or are otherwise unsuitable for MRI-based RT treatment
* Metastatic disease

Ages: 50 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 17 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2034-07-01 (Estimated)

PRIMARY OUTCOMES:
Comparing local recurrence rates between patients receiving Standard CT radiation therapy (ARM1) and MRI-based radiation therapy (ARM 2) | 24months

SECONDARY OUTCOMES:
Comparing local recurrence rates between patients receiving Standard CT radiation therapy (ARM1) and MRI-based radiation therapy (ARM 2) | 60 months
Comparing number of participants with local recurrence between patients treated on Standard CT radiation therapy (ARM1) and MRI-based radiation therapy (ARM 2) | 120 months
Comparing clinical and planning target volumes (CTV and PTV volumes) for CT-based planning vs. MRI-based planning | 60 months
Comparing patient reported cosmetic outcomes between patients treated on Standard CT radiation therapy (ARM1) and MRI-based radiation therapy (ARM 2) | 60 months
  Comparing patient reported cosmetic outcomes between patients treated on Standard CT radiation therapy (ARM1) and MRI-based radiation therapy (ARM 2) using the Breast Cancer Treatment Outcome Scale (BCTOS). BCTOS is a widely used questionnaire that is used to compare outcomes of treated and untreated breast by the patient. The questionnaire includes a cosmetic, functional and breast sensitivity questions.
  BCTOS Cosmesis scores range from 1 (excellent) to 4 (poor), and scores of 3 (fair) or more indicate adverse cosmetic outcomes.
Comparing the number of treatment related acute skin toxicities observed in patients who received either Standard CT radiation therapy (ARM1) and MRI-based radiation therapy (ARM 2) | 6 months
  Comparing the number of treatment related acute skin toxicities observed in patients who received either Standard CT radiation therapy (ARM1) and MRI-based radiation therapy (ARM 2) using the National Cancer Institute Common Toxicity Criteria for Adverse Events, version 5.0 (NCI CTCAEv5.0).
Comparing the number of treatment related acute skin toxicities observed in patients who received either Standard CT radiation therapy (ARM1) and MRI-based radiation therapy (ARM 2) | 12 months
  Comparing the number of treatment related acute skin toxicities observed in patients who received either Standard CT radiation therapy (ARM1) and MRI-based radiation therapy (ARM 2) using the National Cancer Institute Common Toxicity Criteria for Adverse Events, version 5.0 (NCI CTCAEv5.0).
Comparing the number of treatment related acute skin toxicities observed in patients who received either Standard CT radiation therapy (ARM1) and MRI-based radiation therapy (ARM 2) | 24 months
  Comparing the number of treatment related acute skin toxicities observed in patients who received either Standard CT radiation therapy (ARM1) and MRI-based radiation therapy (ARM 2) using the National Cancer Institute Common Toxicity Criteria for Adverse Events, version 5.0 (NCI CTCAEv5.0).
Comparing the number of treatment related late skin toxicities who received either Standard CT radiation therapy (ARM1) and MRI-based radiation therapy (ARM 2) | 6 months
  Comparing the number of treatment related late skin toxicities who received either Standard CT radiation therapy (ARM1) and MRI-based radiation therapy (ARM 2) using the National Cancer Institute Common Toxicity Criteria for Adverse Events, version 5.0 (NCI CTCAEv5.0).
Comparing the number of treatment related late skin toxicities who received either Standard CT radiation therapy (ARM1) and MRI-based radiation therapy (ARM 2) | 12 months
  Comparing the number of treatment related late skin toxicities who received either Standard CT radiation therapy (ARM1) and MRI-based radiation therapy (ARM 2) using the National Cancer Institute Common Toxicity Criteria for Adverse Events, version 5.0 (NCI CTCAEv5.0).
Comparing the number of treatment related late skin toxicities who received either Standard CT radiation therapy (ARM1) and MRI-based radiation therapy (ARM 2) | 24 months
  Comparing the number of treatment related late skin toxicities who received either Standard CT radiation therapy (ARM1) and MRI-based radiation therapy (ARM 2) using the National Cancer Institute Common Toxicity Criteria for Adverse Events, version 5.0 (NCI CTCAEv5.0).

CONTACTS AND LOCATIONS:
Overall Officials: John Ng, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No